CLINICAL TRIAL: NCT01047397
Title: A Phase IIa, Randomized, Single-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of 28-day Repeat Oral Doses of GSK1278863A in Anemic Pre-dialysis and Hemodialysis-dependent Patients
Brief Title: Repeat Dose Safety and Efficacy Study for Compound to Treat Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 112844; PHI112844 (Other: Octagon Research)
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-07

CONDITIONS: Kidney Disease
Keywords: hemodialysis; tolerability; pharmacokinetics; safety; anemia; renal impairment; repeat dose
MeSH Terms: conditions — Kidney Diseases; Anemia; Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Active Drug
  Interventions: Drug: 1278863A
- Group 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 1278863A — 25mg, 50mg, 100mg
  Arms: Group 1
Drug: Placebo — matching placebo
  Arms: Group 2

SUMMARY:
The purpose of this study is to characterize the safety and efficacy of repeat doses of compound 1278863A in subjects with anemia.

DETAILED DESCRIPTION:
Compound 1278863A is a novel small molecule agent, which stimulates erythropoiesis through inhibition of hypoxia-inducible factor (HIF)-prolyl hydroxylases (EGLNs). This compound is being developed for the treatment of anemia. This study, PHI112844, will be the first administration of compound 1278863A to investigate the pharmacodynamics/efficacy, safety, tolerability, and pharmacokinetics of repeat oral doses in anemic pre-dialysis patients with moderate or severe renal impairment and in hemodialysis-dependent patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 85 years of age inclusive, at the time of signing the informed consent.
2. A male or female is eligible to enroll and participate in this study if he/she:

   1. (Part 1) has Moderate to Severe Renal Impairment (equivalent to NKF KDOQI Stage 3 or 4, not receiving dialysis) as determined by estimated Glomerular Filtration Rate (eGFR) calculated by the abbreviated MDRD equation, and not expected to go on dialysis until ≥ 8 weeks after first administration of investigational product. Stage 5, non-dialysis patients with eGFR of 10 15 mL/min per 1.73 m2 will also be eligible for Part 1 on a case-by-case basis.
   2. (Part 2) has Severe Renal Impairment and has been on stable hemodialysis treatment for 1 month prior to Screening (subjects with planned transition to hemodialysis) or 3 months prior to Screening (subjects emergently placed on hemodialysis). These subjects are equivalent to NKF KDOQI Stage 5.
   3. otherwise healthy or considered clinically stable with respect to underlying renal impairment and with respect to underlying/chronic disease as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
   4. has clinical laboratory test results that are considered clinically stable in the opinion of the principal investigator, especially if the clinical abnormality or laboratory parameter is deemed associated with the patient's underlying renal impairment.
3. Meets the following erythropoiesis stimulating agent (ESA) criteria:

   1. The patient is ESA naïve OR
   2. If the patient has a scheduled ESA interval which is ≤ 7 days, ESA treatment must be discontinued for at least 7 days OR
   3. If the patient has a scheduled ESA interval which is > 7 days, ESA treatment must be discontinued for at least that scheduled interval length (eg discontinued ≥ 14 days for a scheduled 14 day ESA interval) AND The patient will not resume ESA treatment until completion of the Follow-up Visit (Day 57).
4. Has a hemoglobin value:

   1. For ESA naïve patients: ≤11.0 g/dL
   2. For patients receiving ongoing ESA treatment: ≤11.5 g/dL at Screening with a re check value of ≤11.0 g/dL after appropriate ESA discontinuation according to Inclusion 3 and prior to commencing study drug dosing.
5. 5. Has serum ferritin at Screening:

   1. ≥40 μg/L with the absence of microcytic or hypochromic RBCs (regardless of transferrin saturation %) OR
   2. 25-39 μg/L with transferrin saturation % ≥20% (fraction saturation ≥0.20) and the absence of microcytic or hypochromic RBCs
6. Has Vitamin B12 and folate above the lower limit of normal at Screening
7. A female patient is eligible to participate if she is:

   1. of childbearing potential, and must agree to use one of the contraception methods in Section 8.1.1. This criterion must be followed from the time of Screening until completion of the Follow-up Visit (Day 57) OR
   2. of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
8. Male patients must agree to use one of the contraception methods listed in Section 8.1.2. This criterion must be followed from the time of the first dose of study drug until completion of the Follow-up Visit (Day 57).
9. Body weight ≥ 45 kg
10. QTcB or QTcF < 450 msec; or QTc < 480 msec in patients with bundle branch block. These should be based on an average of triplicate values obtained at Screening.
11. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months prior to Screening and one of the following:

   * evidence of autoimmune anemia
   * prior anti-viral therapy
   * evidence of liver damage
2. A positive test for HIV antibody.
3. A pre-study drug screen that is positive due to drug use not associated with a current medication prescription. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
4. A value at Screening is greater than 1.5 times the upper limit of reference range for AST, ALT, or direct bilirubin.
5. Hemolysis/hemolytic anemia or active bleeding/blood loss
6. Androgen therapy within 8 weeks prior to first dose of study drug (Day 1).
7. Red blood cell transfusion within 90 days prior to first dose of study drug (Day 1).
8. 8. Iron replacement therapy:

   1. Intravenous iron replacement therapy within 30 days prior to the first dose of study drug on Day 1 until completion of the Follow-up Visit (Day 57).
   2. Oral iron replacement therapy started or discontinued within 30 days prior to Screening. (Patients currently receiving oral iron replacement therapy which was initiated at least 30 days prior to Screening, will be allowed to continue their oral iron replacement therapy during the study and should not discontinue the therapy until after completion of all study drug doses and Day 29 assessments.)
9. History of thrombosis defined as deep vein thrombosis, stroke, pulmonary embolism or other thrombosis related condition within 1 year prior to Screening.
10. Known active decompensated hyperparathyroidism or history of bone marrow fibrosis.
11. Systemic hematologic disease, including, but not limited to sickle cell disease, hemosiderosis, hemochromatosis, myelodysplastic syndrome, hematologic malignancy, myeloma
12. Post-renal transplantation patients with functioning transplant. (Failed transplant subjects back on hemodialysis are eligible).
13. Acute peptic ulcer disease or history of chronic rectal bleeding.
14. History of malignancy tumor within 5 years prior to Screening or are receiving medication for cancer. Non-melanoma skin cancer within the past 5 years that has been definitively removed is allowed.
15. Patients with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, and/or hepatic function that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Examples of conditions that could interfere with normal gastrointestinal anatomy or motility include gastrointestinal bypass surgery, partial or total gastrectomy, small bowel resection, vagotomy, malabsorption, Crohn's disease, ulcerative colitis, or celiac sprue. Examples of conditions that could interfere with hepatic function include Gilberts syndrome.
16. Active infection or acute inflammatory disease as determined by clinical assessment.
17. Class III heart failure with evidence of recent progression (worsening dyspnea, hospitalization within 2-3 months for symptoms, etc), or Class IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system.
18. Uncontrolled hypertension (diastolic BP >100 mmHg or systolic BP >160 mmHg at Screening)
19. Myocardial infarction or acute coronary syndrome within 1 year prior to Screening.
20. History of seizure disorder.
21. Proliferative choroidal or retinal disease, such as neovascular age-related macular degeneration or proliferative diabetic retinopathy that is likely to require treatment (intraocular injections or laser photocoagulation) during the study.
22. Pregnant females as determined by positive serum or urine hCG test at Screening or prior to the first dose of study drug (Day 1).
23. Lactating females.
24. History of drug abuse or dependence within 6 months prior to Screening.
25. Unwillingness or inability to follow the procedures, or lifestyle and/or dietary restrictions outlined in the protocol.
26. Use of prescription drugs within 7 days prior to first dose of study drug (Day 1) until after completion of all study drug doses and Day 29 assessments:

    * which are know to be inhibitors of CYP 2C8 OR
    * which are known to be both CYP 2C8 and OATP1B1 substrates OR
    * which rely mainly on OATP1B1/1B3 for hepatic clearance as described in Section 9 of the protocol.
27. Use of prescription drugs within 14 days prior to first dose of study drug (Day 1) until completion of all study drug doses and Day 29 assessments, which are known to be inducers of CYP 2C8, as described in Section 9 of the protocol.
28. Use of non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study drug (Day 1) through the Follow-up Visit (Day 57), unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise patient safety and GSK Medical Monitor concurs.
29. History of sensitivity to any of the study drugs, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
30. History of sensitivity to heparin or heparin-induced thrombocytopenia. (if the clinical site uses heparin to maintain intravenous cannula patency)
31. The patient has participated in a clinical trial and has received an experimental investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
32. Exposure to more than four experimental investigational products within 12 months prior to the first dose of study drug (Day 1).
33. Patient is mentally or legally incapacitated.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Rate of response for increase from baseline of hemoglobin levels | Pre-dose, Day 1, Day 15, Day 22, Follow-up
Adverse Events reporting | throughout study
Safety Labs (Chemistry) | Screening, Day 1, 4, 8, 15, 22, 29, 36, 57
Safety Labs (Hematology) | Screening, Day 1, 4, 8, 15, 22, 29, 36, 57
Safety Labs (Urinalysis) | Screening, Day 1, 4, 8, 15, 22, 29, 36, 57
Vital Signs (blood pressure and heart rate) | Screening, Day 1, 4, 8, 15, 22, 29, 36, 57
ECG | Screening, Day 1, 4, 8, 15, 22, 29, 36, 57

SECONDARY OUTCOMES:
AUC (0-∞), Cmax, tmax, t½ | Day 1, 15, 22
Actual values and change from baseline for erythropoietin, absolute and percent reticulocytes, hematocrit, and total RBCs | Day 1, 15, 22, Folllow-up
Actual values and change from baseline for VEGF, hepcidin, TIBC | Day 1, 15, 22, Follow-up
Actual values and change from baseline for transferrin saturation, serum iron, serum ferritin | Screening, Day 1, 15, 29, 57
Actual value and change from baseline for fetal hemoglobin | Day 1, 29, 57

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (23):
- Australia (6):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Gosford, New South Wales
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Reservoir, Victoria
- India (6):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Kalapet Pondicherry
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Visakhapatnam
- New Zealand (2):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
- Russia (9):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Volzhsky
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278